CLINICAL TRIAL: NCT00966329
Title: Pilot Study to Assess the Safety and Efficacy of Switching the Nnrti or pi to Maraviroc in Hiv-1-infected Subjects With Persistent Viremia Suppression
Brief Title: Switching the Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI) or Protease Inhibitor (PI) to Maraviroc in HIV Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Sílvia Gel, Dra. Eugenia Negredo, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARAVI-SWITCH
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: HIV; HIV Infections
Keywords: Switching; Maraviroc; Virological efficacy; Lipid profile; Tropism
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- to switch from the NNRTI/PI to maraviroc (Experimental): to switch from the NNRTI/PI to maraviroc
  Interventions: Drug: maraviroc
- to continue with the same approach (Active Comparator): to continue with the same approach
  Interventions: Drug: control group

INTERVENTIONS:
Drug: maraviroc — HAART regimen including 2 NRTI/NtRTIs plus maraviroc
  Arms: to switch from the NNRTI/PI to maraviroc
Drug: control group — HAART regimen including 2 NRTI/NtRTIs plus one of the following :
  * 1 PI/ritonavir (lopinavir/ritonavir, atazanavir/ritonavir, fosamprenavir /ritonavir, tipranavir/ritonavir, darunavir/ritonavir)
  * or ATV/unboosted (in a regimen without tenofovir)
  * or 1 NNRTI (nevirapine or efavirenz).
  Arms: to continue with the same approach

SUMMARY:
Patients with HIV-1 infection on HAART regimen including 2 NRTI/NtRTIs plus one of the following : 1 PI/ritonavir or ATV/unboosted or 1 NNRTI, will be randomized to switch from the NNRTI/PI to maraviroc (300 mg /12 h) or to continue with the same approach.

DETAILED DESCRIPTION:
This is a 48 week randomized, prospective, controlled, open-label, proof-of-concept pilot clinical trial.

Patients with HIV-1 infection on HAART regimen including 2 NRTI/NtRTIs plus one of the following : 1 PI/ritonavir (lopinavir/ritonavir, atazanavir/ritonavir, fosamprenavir /ritonavir, tipranavir/ritonavir, darunavir/ritonavir) or ATV/unboosted (in a regimen without tenofovir) or 1 NNRTI (nevirapine or efavirenz).

Patients will be randomized to switch from the NNRTI/PI to maraviroc (300 mg /12 h) or to continue with the same approach.

The primary endpoint would be the percentage of patients who maintain virological suppression at week 48.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected adults (=/+18 years old).
2. Patient having a diagnosis of HIV infection, on stable HAART including 2 NRTI/NtRTIs plus one of the following: 1 PI/ritonavir or ATV/unboosted or 1 NNRTI.
3. Undetectable plasma HIV-1 RNA (VL < 50 copies/mL) while on HAART.
4. Patient having at least one of the following conditions:

   * Antiretroviral-related gastrointestinal disturbances, or
   * Low patient's satisfaction associated with the current regimen posology (ritonavir use, ritonavir intolerance…), or
   * Any toxicity drug related.
5. Nadir CD4 cell count > 350 cells/mm3.
6. Absence of resistance mutations in the RT or PR by (TrugeneTM)
7. Good treatment adherence.
8. Voluntary written informed consent.

Exclusion Criteria:

1. Virologic failure to a previous antiretroviral regimen.
2. Any antiretroviral resistance mutation in a previous resistance test.
3. Dual/mixed or X4 viruses detected at any time point, including the pre-treatment ES-Trofile test of the PBMC test done before treatment switch.
4. Acute infections or uncontrolled chronic infection in the 2 months previous to the inclusion.
5. Pregnancy or fertile women willing to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Viral load | 48 weeks

SECONDARY OUTCOMES:
Time to virological failure | 48 weeks
Administration of lipid-lowering drugs | 48 weeks
Changes in the SCORE equation | 48 weeks
CD4 / CD8 cell counts | 48 weeks
Antiretroviral resistance and viral tropism | 48 weeks
Patients who withdraw | 48 weeks
Total cholesterol | 48 weeks
  Total cholesterol levels
HDL-cholesterol | 48 weeks
  HDL-cholesterol levels
LDL-cholesterol | 48 weeks
  LDL-cholesterol levels
Triglyceride | 48 weeks
  Triglyceride levels

CONTACTS AND LOCATIONS:
Overall Officials: Eugènia Negredo, MD,PhD, Principal Investigator — Lluita contra la Sida Foundation, HIV Unit
Locations (3):
- Spain (3):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Lluita contra la Sida Foundation, HIV Unit, Irsi Caixa Foundation, Badalona, Barcelona
  - Lluita contra la Sida Foundation, HIV Unit, Badalona, Barcelona

REFERENCES:
- [Derived] Bonjoch A, Pou C, Perez-Alvarez N, Bellido R, Casadella M, Puig J, Noguera-Julian M, Clotet B, Negredo E, Paredes R. Switching the third drug of antiretroviral therapy to maraviroc in aviraemic subjects: a pilot, prospective, randomized clinical trial. J Antimicrob Chemother. 2013 Jun;68(6):1382-7. doi: 10.1093/jac/dks539. Epub 2013 Jan 25. PMID 23354282